CLINICAL TRIAL: NCT00603733
Title: A Multicentre, Randomised, Double-blind, Non-inferiority Trial Comparing the Efficacy and Safety of a New Modified Oral Extended Release Pentasa® (Mesalamine) 500 mg Tablet to the Currently Marketed Pentasa® (Mesalamine) 500 mg Tablet in Subjects With Active Mild to Moderate Ulcerative Colitis Treated With 4 g/Day for 8 Weeks and in Maintenance of Remission of Ulcerative Colitis in Subjects Treated With 2 g/Day for 24 Weeks
Brief Title: Canadian Active & Maintenance Modified Pentasa Study
Acronym: CAMMP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLN 35.3.11
Record Dates: First submitted 2008-01-16; First posted 2008-01-29 (Estimated); Results first posted 2016-04-22 (Estimated); Last update posted 2016-04-22 (Estimated); Status verified 2016-04

CONDITIONS: Active Ulcerative Colitis; Remission of Ulcerative Colitis
Keywords: Ulcerative Colitis; 5-Aminosalicylate
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Mesalamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pentasa® modified extended release (Experimental): 5-ASA (5-Aminosalicylate)
  Interventions: Drug: 5-ASA (5-Aminosalicylate)
- Pentasa® (Active Comparator): 5-ASA (5-Aminosalicylate)
  Interventions: Drug: 5-ASA (5-Aminosalicylate)

INTERVENTIONS:
Drug: 5-ASA (5-Aminosalicylate) — 500 mg tablet (modified extended release)
  Other Names: Pentasa®; mesalamine
  Arms: Pentasa® modified extended release
Drug: 5-ASA (5-Aminosalicylate) — 500 mg tablet
  Other Names: Pentasa®; mesalamine
  Arms: Pentasa®

SUMMARY:
The purpose of this study is to demonstrate that the new modified oral extended-release Pentasa® 500mg tablet is at least as efficacious as the currently marketed Pentasa® 500mg tablet in active mild to moderate Ulcerative Colitis (UC) and also in maintenance of quiescent disease.

DETAILED DESCRIPTION:
A multi-centre, randomized, double-blind, non-inferiority trial comparing the efficacy and safety of a new modified oral extended release Pentasa® (mesalamine) 500 mg tablet to the currently marketed Pentasa® (mesalamine) 500 mg tablet in subjects with active mild to moderate ulcerative colitis treated with 4 g/day for 8 weeks and in maintenance of remission of ulcerative colitis in subjects treated with 2 g/day for 24 weeks. The study involves male or non-pregnant female subjects aged 18 to 75 years.

Subjects were randomised on entry into the trial, and if they were in remission at the end of the 8-week Active Phase or the 4-week Run-in Phase, they were eligible for enrolment into the 24-week Maintenance Phase, remaining on the original randomised treatment.

ELIGIBILITY:
Inclusion Criteria for Active phase:

* Newly diagnosed or recurrent, mild to moderate Ulcerative Colitis patients.
* Extent of colonic involvement confirmed within the past 36 months
* UCDAI score of at least 3 but not greater than 8 and a score of at least 1 for endoscopy
* Screening tests to rule out any abnormalities in stool, heart or kidney.
* Male or non-pregnant females between 18 to 75 years.
* Women of childbearing potential to use efficacious contraception as judged by the investigator.
* Written informed consent given.

Inclusion Criteria for Maintenance phase:

* Newly recruited subjects with documented mild to moderate UC entering the Run-in Phase: in clinical remission for at least 1 month and for a maximum of 3 years, and receiving 5-ASA 1.4 to 2.5 g/day for maintenance of quiescent disease
* Subjects from Active Phase: meeting remission criteria after the 8-week active period
* Extent of colonic involvement confirmed within the past 36 months by colonoscopy
* In complete remission at entry into the Maintenance Phase, defined as i) a score of 0 or 1 for stool frequency; ii) a score of 0 for rectal bleeding; iii) a score of 0 for endoscopy findings; and iv) a Physician's Global Assessment (PGA) score of 0 or 1
* Screening tests to rule out any abnormalities in stool, heart or kidney.

Exclusion Criteria:

* Use of 5-ASA products at a dose >2.5g/day within 7 days prior to entry.
* Proctitis, short bowel syndrome, prior bowel surgery, severe UC, other forms of Inflammatory Bowel Disease
* Infectious diseases, parasites, bacterial pathogens
* Allergy to aspirin or salicylate
* Liver or kidney abnormalities
* Alcohol or drug abuse
* Pregnancy
* Cancer
* Bleeding disorders, ulcers, autoimmune diseases
* Mental disorders
* Participation in clinical trial in last 30 days
* Inability to fill in diary cards / comply with protocol requirements

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Actual)
Dates: Start 2007-10; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (27):
- Canada (27):
  - University of Calgary, Faculty of Medicine, Calgary, Alberta
  - Castledowns Medicentre, Edmonton, Alberta
  - Investigational site, Brandon, Manitoba
  - Hilyard Place Building A, Saint John, New Brunswick
  - Barrie GI Associates, Barrie, Ontario
  - Investigational site, Greater Sudbury, Ontario
  - Investigational site, Guelph, Ontario
  - St. Joseph's Healthcare, Hamilton, Ontario
  - Investigational site, Oshawa, Ontario
  - Investigational site - Phenix Building, Ottawa, Ontario
  - Ottawa General Hospital, Ottawa, Ontario
  - Digestive Health Clinic, Richmond Hill, Ontario
  - Investigational site, Sarnia, Ontario
  - Investigational site, Thunder Bay, Ontario
  - JJ Dig Research Ltd, Toronto, Ontario
  - Keele Medical Place, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Toronto Digestive Disease Association (TDDA), Toronto, Ontario
  - Hotel Dieu Grace Hospital, Windsor, Ontario
  - Investigational site, Windsor, Ontario
  - Investigational site, Woodstock, Ontario
  - Hotel Dieu de Levis, Lévis, Quebec
  - Alpha Recherche Clinique Inc., Loretteville, Quebec
  - Hopital Maissonneuve Rosemont, Montreal, Quebec
  - MUHC-Royal Victoria Hospital, Montreal, Quebec
  - Gastro Centre Hospitalier Universitaire de Québec/St-François-d'Assise Hospital, Québec, Quebec
  - L'Hotel Dieu de Quebec, Québec, Quebec

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Total number of unique patients enrolled in the study is 288 whereby 190 patients were enrolled in the Active Phase and 98 patients were enrolled in the Run-In Phase.
  The patients enrolled in the Maintenance Phase are a combination of patients who completed the Active (82) and Run In (71) Phases and were eligible to move forward into Maintenance.
Period: Active Phase ITT
Arm/Group | Pentasa® Modified Extended Release | Pentasa®
Started | 95 (Note: a total of 190 new participants were enrolled and randomized in the Active Phase) | 95
Completed | 84 | 78
Not Completed | 11 | 17
Not completed — Adverse Event | 8 | 7
Not completed — Withdrawal by Subject | 0 | 3
Not completed — Lost to Follow-up | 0 | 1
Not completed — Did not meet inclusion/exclusion | 1 | 3
Not completed — Lack of Efficacy | 1 | 2
Not completed — Subject moved, site closed | 1 | 1
Period: Run-In Phase - 4 Weeks
Arm/Group | Pentasa® Modified Extended Release | Pentasa®
Started | 49 (Note: Of the 98 subjects randomized at Run-In, 71 progressed into the maintenance phase.) | 49
Completed | 35 | 36
Not Completed | 14 | 13
Not completed — Adverse Event | 2 | 1
Not completed — Withdrawal by Subject | 4 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Did not meet incl/excl criteria | 5 | 10
Not completed — Lack of Efficacy | 2 | 1
Period: Maintenance Phase ITT
Arm/Group | Pentasa® Modified Extended Release | Pentasa®
Started | 71 (Note:82 subjects randomized at Active phase & 71 at Run-In phase progressed to the maintenance phase) | 82
Completed | 61 | 66
Not Completed | 10 | 16
Not completed — Adverse Event | 3 | 6
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Protocol Violation | 1 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Lack of Efficacy | 2 | 2
Not completed — Physician Decision | 0 | 1
Not completed — Site withdrew, subject away, lost IMP | 3 | 5

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were reported for the Per Protocol population who participated in the Active phase and in the maintenance phase of this study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pentasa® Modified Extended Release | Pentasa® | Total
Number analyzed (Participants) | 139 | 146 | 285
Age, Continuous [Mean (Standard Deviation); unit: years]
  Active Phase | 44.2 (12.88) | 44.5 (12.53) | 44.35 (12.71)
  Maintenance Phase | 46.4 (12.20) | 45.8 (13.45) | 46.1 (12.83)
Age, Customized [Median (Full Range); unit: years]
  Active Phase | 45 [18 to 68] | 43.5 [22 to 76] | 44.3 [18 to 76]
  Maintenance Phase | 48 [20 to 65] | 44.5 [23 to 76] | 46.3 [20 to 76]
Sex/Gender, Customized [Number; unit: participants]
  Active Phase, Female | 30 | 34 | 64
  Active Phase, Male | 48 | 44 | 92
  Maintenance Phase, Female | 28 | 29 | 57
  Maintenance Phase, Male | 33 | 39 | 72
Region of Enrollment [Number; unit: participants]
  Canada | 139 | 146 | 285

OUTCOME MEASURES:

1. Primary Outcome: Active Phase: Proportion of Active Subjects Achieving Overall Improvement
Description: Overall improvement is defined as either a complete remission or a clinical response to therapy as measured by the Ulcerative Colitis Disease Activity Index (UCDAI).
  Complete remission is defined as: i) a score of 0 or 1 for stool frequency; ii) a score of 0 for rectal bleeding; iii) a score of 0 for endoscopy findings and iv) a Physician's Global Assessment (PGA) score of 0 or 1.
  A clinical response to therapy in the active disease phase is defined as i) improvement in the baseline PGA score; ii) improvement in endoscopy findings and in at least one other clinical assessment (stool frequency, rectal bleeding); iii) no worsening in any other clinical assessment; iv) a decrease of 2 or more points on the UCDAI score.
Time Frame: From baseline to week 8
Population: Per Protocol Analysis Set
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Pentasa® Modified Extended Release | Pentasa®
Number analyzed (Participants) | 78 | 78
percentage of participants | 64.1 [55.17 to 73.04] | 69.2 [60.63 to 77.83]

2. Primary Outcome: Maintenance Phase: Proportion of Subjects Experiencing Relapse
Description: Relapse is defined as a UCDAI score of at least 3 and a score of at least 1 for endoscopy
Time Frame: Up to week 24
Population: Per Protocol Analysis Set
Measure: Number (90% Confidence Interval); unit: % of subjects with relapse (90% CI)
Arm/Group | Pentasa® Modified Extended Release | Pentasa®
Number analyzed (Participants) | 61 | 68
% of subjects with relapse (90% CI) | 24.6 [15.52 to 33.66] | 11.8 [5.34 to 18.19]

3. Secondary Outcome: Frequency of Adverse Events
Description: Safety dataset represents all patients in all study phases exposed to study drug at anytime during study. Safety dataset was a combination of the active, run-in and maintenance phases and therefore it is not possible to report the adverse events per phase.
Time Frame: From baseline to week 24
Population: Safety dataset for Active and Maintenance Phases
Measure: Number; unit: percentage of patients with TEAEs
Arm/Group | Pentasa® Modified Extended Release | Pentasa®
Number analyzed (Participants) | 143 | 144
percentage of patients with TEAEs | 52.4 | 45.1

ADVERSE EVENTS:
Time Frame: Adverse Event data is collected from the time Informed Consent is taken up to 28 days post study.
Description: Safety dataset represents all patients in all study phases exposed to study drug at anytime during study. Safety dataset was a combination of the active, run-in and maintenance phases and therefore it is not possible to report the adverse events per phase.
Arm/Group | Pentasa® Modified Extended Release | Pentasa®
Serious Adverse Events (participants affected / at risk) | 7/143 | 2/144
Other Adverse Events (participants affected / at risk) | 27/143 | 28/144
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pentasa® Modified Extended Release (N=143) | Pentasa® (N=144)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pentasa® Modified Extended Release (N=143) | Pentasa® (N=144)
Colitis Ulcerative (Gastrointestinal disorders) | 4 (4) | 9 (10)
Nasopharyngitis (Infections and infestations) | 12 (15) | 6 (8)
Headache (Nervous system disorders) | 11 (12) | 13 (15)

LIMITATIONS AND CAVEATS:
Study was amended to modify sample size as subject enrolment was lower than anticipated. A data lock was imposed, pending completion of the Maintenance Phase by 12 subjects to report all Active Phase efficacy data & all available safety data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review the draft manuscript prior to publication and can request delay of publication where any contents are deemed patentable by the sponsor or confidential to the sponsor. Comments will be given within four weeks from receipt of the draft manuscript. Additional time may be required to allow Ferring to seek patent protection of the invention.